CLINICAL TRIAL: NCT03321968
Title: A Randomized, Observer-blind, Multicenter, Phase 3 Study to Evaluate the Lot Consistency, Immunogenicity, and Safety of a Plant-Derived Quadrivalent VLP Influenza Vaccine in Healthy Adults 18-49 Years of Age
Brief Title: Lot-to-lot Consistency of a Plant-Derived Quadrivalent Virus-Like Particles Influenza Vaccine in Healthy Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medicago (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CP-PRO-QVLP-011
Record Dates: First submitted 2017-10-16; First posted 2017-10-26 (Actual); Results first posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Virus Diseases; RNA Virus Infections; Respiratory Tract Infections; Respiratory Tract Disease; Influenza
Keywords: Influenza; Human; RNA Virus Infections; Lot Consistency; Immunologic; Orthomyxoviridae Infections; Infection; Virus Diseases; Vaccine; Safety; Plant-made; Virus-like particle; Hemagglutinin
MeSH Terms: conditions — Virus Diseases; RNA Virus Infections; Respiratory Tract Infections; Respiratory Tract Diseases; Influenza, Human; Orthomyxoviridae Infections; Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Quadrivalent VLP Influenza Vaccine - Lot 1 (Experimental): Participants received one intramuscular (IM) injection of 0.5 mL of their assigned vaccine lot of 30 μg/strain of the Quadrivalent VLP Influenza Vaccine on Day 0.
  Interventions: Biological: Quadrivalent VLP Influenza Vaccine
- Quadrivalent VLP Influenza Vaccine - Lot 2 (Experimental): Participants received one IM injection of 0.5 mL of their assigned vaccine lot of 30 μg/strain of the Quadrivalent VLP Influenza Vaccine on Day 0.
  Interventions: Biological: Quadrivalent VLP Influenza Vaccine
- Quadrivalent VLP Influenza Vaccine - Lot 3 (Experimental): Participants received one IM injection of 0.5 mL of their assigned vaccine lot of 30 μg/strain of the Quadrivalent VLP Influenza Vaccine on Day 0.
  Interventions: Biological: Quadrivalent VLP Influenza Vaccine

INTERVENTIONS:
Biological: Quadrivalent VLP Influenza Vaccine — Single dose of 30 µg/strain Quadrivalent VLP Influenza Vaccine

SUMMARY:
This Phase 3 study is intended to assess the clinical lot-to-lot consistency in manufacturing by evaluating and comparing the immunogenicity of three consecutively manufactured lots of the Quadrivalent Virus-Like Particles (VLP) Influenza Vaccine, during the 2016-2017 influenza season, in healthy adults 18-49 years of age. A single dose of one of three consecutive lots of Quadrivalent VLP Influenza Vaccine (30 µg/strain) will be administered to 1,200 participants.

DETAILED DESCRIPTION:
This randomized, observer-blind, multicenter, Phase 3 lot consistency study will be conducted at multiple sites in Canada. The composition of the Quadrivalent VLP Influenza Vaccine used in this study includes two influenza A virus strains and two influenza B virus strains based on the 2016-2017 recommended strains for vaccination in the Northern hemisphere.

1,200 healthy male and female participants aged 18 to 49 years will be randomized in a 1:1:1 ratio to one of three lots of the Quadrivalent VLP Influenza Vaccine (30 μg/strain). Participant will participate in this study for approximately 21 days, during which a first visit will be scheduled on Day 0 for screening, eligibility assessment, and vaccine administration; and on Day 21 for blood sample collection for immunogenicity assessment.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following inclusion criteria to be eligible for participation in this study; no protocol waivers are allowed:

1. Participants must be considered by the Investigator to be reliable and likely to cooperate with the assessment procedures and be available for the duration of the study;
2. Participants have a body mass index (BMI) ≤ 40.0 kg/m^2 on Day 0 (pre-vaccination);
3. Participants must be in good general health prior to study participation with no clinically relevant abnormalities that could jeopardize participant safety or interfere with study assessments as assessed by the Principal Investigator or sub-Investigator (thereafter referred as Investigator) and determined by medical history, physical examination, and vital signs; Note: Participants with a pre-existing chronic disease will be allowed to participate if the disease is stable and, according to the Investigator's judgment, the condition is unlikely to confound the results of the study or pose additional risk to the participant by participating in the study. Stable disease is generally defined as no new onset or exacerbation of pre-existing chronic disease six months prior to vaccination. Based on the Investigator's judgment, a participant with a more recent stabilization of a disease could also be eligible.
4. Female participants must have a negative urine pregnancy test result at the Screening/Vaccination visit (Visit 1);
5. Female participants of childbearing potential must use an effective method of contraception for one month prior to vaccination and agree to continue employing adequate birth control measures for the duration of the study. Abstinent participants should be asked what method(s) they would use, should their circumstances change, and participants without a well-defined plan should be excluded. The following relationship or methods of contraception are considered to be effective:

   * Hormonal contraceptives (e.g. oral, injectable, topical [patch], or estrogenic vaginal ring);
   * Intra-uterine device with or without hormonal release;
   * Male partner using a condom plus spermicide or a sterilized partner (at least one year prior to vaccination);
   * Credible self-reported history of heterosexual vaginal intercourse abstinence until at least the Day 21 visit;
   * Female partner.
6. Non-childbearing females are defined as:

   * Surgically-sterile (defined as bilateral tubal ligation, hysterectomy, or bilateral oophorectomy performed more than one month prior to vaccination); or
   * Post-menopausal (absence of menses for 24 consecutive months and age consistent with natural cessation of ovulation).

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from participating in this study; no protocol waivers are allowed:

1. According to the Investigator's opinion, history of significant acute or chronic, uncontrolled medical or neuropsychiatric illness. 'Uncontrolled' is defined as:

   * Requiring a new medical or surgical treatment during the six months prior to study vaccine administration unless the criteria outlined in inclusion criterion no. 3 can be met (i.e. the Investigator can justify inclusion based upon the innocuous nature of medical/surgical events and/or treatments);
   * Requiring any significant change in a chronic medication (i.e. drug, dose, frequency) during the three months prior to study vaccine administration due to uncontrolled symptoms or drug toxicity, unless the innocuous nature of the medication change meets the criteria outlined in inclusion criterion no. 5 and is appropriately justified by the Investigator.
2. Any medical or neuropsychiatric condition or any history of excessive alcohol use or drug abuse which, in the Investigator's opinion, would render the participant unable to provide informed consent or unable to provide valid safety observations and reporting;
3. Any autoimmune disease other than hypothyroidism with stable replacement therapy; or any confirmed or suspected immunosuppressive condition or immunodeficiency including known or suspected human immunodeficiency virus (HIV), hepatitis B or C infection, or the presence of lymphoproliferative disease;
4. Administration or planned administration of any non-influenza vaccine within 30 days prior to randomization and up to blood sampling on Day 21. Immunization on an emergency basis will be evaluated case-by-case by the Investigator;
5. Administration of any adjuvanted or investigational influenza vaccine within 24 months prior to randomization or planned administration prior to the completion of Day 21;
6. Administration of any "standard", non-adjuvanted influenza vaccine (e.g. live attenuated trivalent/quadrivalent inactivated influenza vaccine intranasal or split trivalent/quadrivalent inactivated influenza vaccine by either intradermal or IM route) within 24 months prior to randomization and up to completion of the Day 21 visit;
7. Use of any investigational or non-registered product within 30 days prior to randomization or planned use during the study period. Participants may not participate in any other investigational or marketed drug study while participating in this study until the Day 21 visit. Participation in observational studies is permitted;
8. Treatment with systemic glucocorticoids at a dose exceeding 10 milligrams (mg) of prednisone (or the equivalent) per day for more than seven consecutive days or for ten or more days in total, within one month of study vaccine administration; or any other cytotoxic or immunosuppressant drug, or any immunoglobulin preparation within three months of vaccination and until the completion of the Day 21 visit. Low doses of nasal or inhaled glucocorticoids and topical steroids are permitted;
9. Any significant disorder of coagulation including, but not limited to, treatment with warfarin derivatives or heparin. Persons receiving prophylactic anti-platelet medications (e.g. low-dose aspirin [no more than 325 mg/day]) and without a clinically apparent bleeding tendency are eligible. Participants treated with new generation drugs that do not increase the risk of IM bleeding (e.g. clopidogrel) are also eligible.
10. History of allergy to any of the constituents of the Quadrivalent VLP Influenza Vaccine or a tobacco allergy;
11. History of anaphylactic allergic reactions to plants or plants components;
12. Any history of serious asthma (e.g. status asthmaticus, hospitalization for asthma control) in the last three years;
13. Use of antihistamines 48 hours prior to study vaccination;
14. The use of prophylactic medications (e.g. acetaminophen/paracetamol, aspirin, naproxen, or ibuprofen) within 24 hours of randomization to prevent or pre-empt symptoms due to vaccination. Participant discovered to have taken a prophylactic medication to prevent or pre empt symptoms due to vaccination within the 24 hours prior to planned randomization must be delayed until at least the 24-hour period is met;
15. Participants who have a dermatological condition at the injection site that may interfere with injection site reaction rating;
16. Participant who have received a blood transfusion within 90 days prior to study vaccination;
17. Any female participant who has a positive or doubtful pregnancy test result prior to vaccination or who is lactating;
18. Presence of any febrile illness (including oral temperature (OT) ≥ 38.0 ˚C within 24 hours prior to vaccination). Such participants may be re-evaluated for enrolment after resolution of illness;
19. Cancer or treatment for cancer within three years of study vaccine administration. Participants with a history of cancer who are disease-free without treatment for three years or more are eligible. Individuals with treated and uncomplicated basal cell carcinoma of the skin or with non-treated, non-disseminated local prostate cancer are eligible;
20. Participants identified as an Investigator or employee of the Investigator or clinical site with direct involvement in the proposed study, or identified as an immediate family member (i.e. parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study or any employee of Medicago. Immediate family members of the Investigator or employees of a clinical site can participate in the study at another clinical site, as long as the Investigator or employees are not involved in the study at that site;
21. Participant with a history of Guillain-Barré syndrome.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1202 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Medicago
Locations (10):
- Canada (10):
  - Site 205, Halifax, Nova Scotia
  - Site 208, Burlington, Ontario
  - Site 207, Guelph, Ontario
  - Site 202, Toronto, Ontario
  - Site 204, Chicoutimi, Quebec
  - Site 203, Gatineau, Quebec
  - Site 201, Lévis, Quebec
  - Site 209, Pointe-Claire, Quebec
  - Site 206, Toronto, Quebec
  - Site 210, Victoriaville, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ward BJ, Seguin A, Couillard J, Trepanier S, Landry N. Phase III: Randomized observer-blind trial to evaluate lot-to-lot consistency of a new plant-derived quadrivalent virus like particle influenza vaccine in adults 18-49 years of age. Vaccine. 2021 Mar 5;39(10):1528-1533. doi: 10.1016/j.vaccine.2021.01.004. Epub 2021 Feb 10. PMID 33581920

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized in a 1:1:1 ratio to receive one of the three lots of the Quadrivalent Virus-Like Particles (VLP) Influenza Vaccine at a dose of 30 μg/strain.
Pre-assignment Details: Participants were healthy adults 18 to 49 years of age assessed during the 2016-2017 influenza season.
Period: Overall Study
Arm/Group | Quadrivalent VLP Influenza Vaccine - Lot 1 | Quadrivalent VLP Influenza Vaccine - Lot 2 | Quadrivalent VLP Influenza Vaccine - Lot 3
Started | 401 | 399 | 402
Vaccinated | 401 | 398 | 401
Completed | 398 | 397 | 399
Not Completed | 3 | 2 | 3
Not completed — Withdrawal by Subject | 1 | 2 | 1
Not completed — Lost to Follow-up | 2 | 0 | 1
Not completed — Other than specified | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set (SAS) was defined as all participants who received Quadrivalent VLP Influenza Vaccine.
Groups:
- Quadrivalent VLP Influenza Vaccine - Lot 1; Quadrivalent VLP Influenza Vaccine - Lot 2; Quadrivalent VLP Influenza Vaccine - Lot 3: Participants received one IM injection of 0.5 mL of their assigned vaccine lot of 30 μg/strain of the Quadrivalent VLP Influenza Vaccine on Day 0.
- Total: Total of all reporting groups
Arm/Group | Quadrivalent VLP Influenza Vaccine - Lot 1 | Quadrivalent VLP Influenza Vaccine - Lot 2 | Quadrivalent VLP Influenza Vaccine - Lot 3 | Total
Number analyzed (Participants) | 401 | 398 | 401 | 1200
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (9.31) | 29.9 (8.90) | 29.4 (8.80) | 29.9 (9.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216 | 224 | 217 | 657
  Male | 185 | 174 | 184 | 543
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 20 | 27 | 68
  Not Hispanic or Latino | 380 | 377 | 374 | 1131
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 63 | 66 | 58 | 187
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 2 | 3
  Black or African American | 17 | 24 | 28 | 69
  White | 318 | 305 | 310 | 933
  More than one race | 2 | 1 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Hemagglutination Inhibition (HI) Antibody Response for Each Homologous Influenza Strain
Description: The GMTs were measured using a HI assay for the homologous strains: A/California/7/2009 (H1N1), A/Hong Kong/4801/2014 (H3N2), B/Brisbane/60/2008 (Victoria lineage), and B/Phuket/3073/2013 (Yamagata lineage). Lot-to-lot consistency was based on adjusted GMT ratio for pairwise comparisons of the lots (Lot 1 / Lot 2, Lot 1 / Lot 3, and Lot 2 / Lot 3).
Time Frame: Day 21 (post-vaccination)
Population: The Per Protocol (PP) analysis set consisted of the participants with no major deviations related to the analyses and with Day 0 and Day 21 immunogenicity assessments.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Quadrivalent VLP Influenza Vaccine - Lot 1 | Quadrivalent VLP Influenza Vaccine - Lot 2 | Quadrivalent VLP Influenza Vaccine - Lot 3
Number analyzed (Participants) | 386 | 383 | 387
titers
  A/H1N1 (California) | 603.7 [541.4 to 673.2] | 595.6 [533.9 to 664.4] | 630.6 [565.6 to 703.0]
  A/H3N2 (Hong Kong) | 96.3 [84.2 to 110.1] | 103.0 [90.0 to 117.7] | 88.0 [77.0 to 100.6]
  B/Brisbane | 41.8 [37.8 to 46.1] | 41.9 [38.0 to 46.3] | 38.3 [34.7 to 42.3]
  B/Phuket | 215.7 [193.2 to 240.9] | 231.1 [206.8 to 258.1] | 235.9 [211.3 to 263.4]
Statistical Analysis 1: Comparison: Quadrivalent VLP Influenza Vaccine - Lot 1 vs Quadrivalent VLP Influenza Vaccine - Lot 2; A/H1N1 (California); Test type: Superiority; Adjusted GMT Ratio = 1.01, 95% CI 2-sided [0.87 to 1.18] — Adjusted GMT/GMT Ratio based on analysis of covariance (ANCOVA) model with vaccine lot as main effect and the baseline titer (log-transformed) as covariate
Statistical Analysis 2: Comparison: Quadrivalent VLP Influenza Vaccine - Lot 1 vs Quadrivalent VLP Influenza Vaccine - Lot 3; A/H1N1 (California); Test type: Superiority; Adjusted GMT Ratio = 0.96, 95% CI 2-sided [0.82 to 1.12] — Adjusted GMT/GMT Ratio based on ANCOVA model with vaccine lot as main effect and the baseline titer (log-transformed) as covariate
Statistical Analysis 3: Comparison: Quadrivalent VLP Influenza Vaccine - Lot 2 vs Quadrivalent VLP Influenza Vaccine - Lot 3; A/H1N1 (California); Test type: Superiority; Adjusted GMT Ratio = 0.94, 95% CI 2-sided [0.81 to 1.10] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Quadrivalent VLP Influenza Vaccine - Lot 1 vs Quadrivalent VLP Influenza Vaccine - Lot 2; A/H3N2 (Hong Kong); Test type: Superiority; Adjusted GMT Ratio = 0.94, 95% CI 2-sided [0.77 to 1.13] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Quadrivalent VLP Influenza Vaccine - Lot 1 vs Quadrivalent VLP Influenza Vaccine - Lot 3; A/H3N2 (Hong Kong); Test type: Superiority; Adjusted GMT Ratio = 1.09, 95% CI 2-sided [0.91 to 1.32] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Quadrivalent VLP Influenza Vaccine - Lot 2 vs Quadrivalent VLP Influenza Vaccine - Lot 3; A/H3N2 (Hong Kong); Test type: Superiority; Adjusted GMT Ratio = 1.17, 95% CI 2-sided [0.97 to 1.41] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Quadrivalent VLP Influenza Vaccine - Lot 1 vs Quadrivalent VLP Influenza Vaccine - Lot 2; B/Brisbane; Test type: Superiority; Adjusted GMT Ratio = 1.00, 95% CI 2-sided [0.87 to 1.15] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: Quadrivalent VLP Influenza Vaccine - Lot 1 vs Quadrivalent VLP Influenza Vaccine - Lot 3; B/Brisbane; Test type: Superiority; Adjusted GMT Ratio = 1.09, 95% CI 2-sided [0.95 to 1.26] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Quadrivalent VLP Influenza Vaccine - Lot 2 vs Quadrivalent VLP Influenza Vaccine - Lot 3; B/Brisbane; Test type: Superiority; Adjusted GMT Ratio = 1.10, 95% CI 2-sided [0.95 to 1.26] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 10: Comparison: Quadrivalent VLP Influenza Vaccine - Lot 1 vs Quadrivalent VLP Influenza Vaccine - Lot 2; B/Phuket; Test type: Superiority; Adjusted GMT Ratio = 0.93, 95% CI 2-sided [0.80 to 1.09] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Quadrivalent VLP Influenza Vaccine - Lot 1 vs Quadrivalent VLP Influenza Vaccine - Lot 3; B/Phuket; Test type: Superiority; Adjusted GMT Ratio = 0.91, 95% CI 2-sided [0.78 to 1.07] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 12: Comparison: Quadrivalent VLP Influenza Vaccine - Lot 2 vs Quadrivalent VLP Influenza Vaccine - Lot 3; B/Phuket; Test type: Superiority; Adjusted GMT Ratio = 0.98, 95% CI 2-sided [0.84 to 1.15] — [estimate comment as in outcome 1, analysis 2]

2. Secondary Outcome: Percentage of Participants With Seroconversion (SC) Measured by HI Antibody Response for Each Homologous Influenza Strain
Description: The SC rate is the percentage of participants with either a ≥ 4-fold increase in reciprocal HI titers between Day 0 and Day 21 or a rise of undetectable HI titer (i.e. <10) pre-vaccination (Day 0) to an HI titer of ≥40 on Day 21 post-vaccination. SC rate was measured using an HI assay for the homologous strains: A/California/7/2009 (H1N1), A/Hong Kong/4801/2014 (H3N2), B/Brisbane/60/2008 (Victoria lineage), and B/Phuket/3073/2013 (Yamagata lineage).
Time Frame: Day 0 (pre-vaccination) to Day 21
Population: PP Set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Quadrivalent VLP Influenza Vaccine - Lot 1 | Quadrivalent VLP Influenza Vaccine - Lot 2 | Quadrivalent VLP Influenza Vaccine - Lot 3
Number analyzed (Participants) | 386 | 383 | 387
percentage of participants
  A/H1N1 (California) | 73.3 [68.6 to 77.7] | 68.7 [63.8 to 73.3] | 73.1 [68.4 to 77.5]
  A/H3N2 (Hong Kong) | 60.9 [55.8 to 65.8] | 63.2 [58.1 to 68.0] | 57.4 [52.3 to 62.4]
  B/Brisbane | 41.2 [36.2 to 46.3] | 42.8 [37.8 to 48.0] | 39.0 [34.1 to 44.1]
  B/Phuket | 63.2 [58.2 to 68.0] | 55.4 [50.2 to 60.4] | 61.2 [56.2 to 66.1]

3. Secondary Outcome: Percentage of Participants With Seroprotection (SP) Measured by HI Antibody Response of for Each Homologous Influenza Strain
Description: The SP rate is the percentage of participants attaining a reciprocal HI titer of ≥ 40 on Day 21 (the percentage of vaccine recipients with a serum HI titer of at least 1:40 following vaccination). SP rate was measured using an HI assay for the homologous strains: A/California/7/2009 (H1N1), A/Hong Kong/4801/2014 (H3N2), B/Brisbane/60/2008 (Victoria lineage), and B/Phuket/3073/2013 (Yamagata lineage).
Time Frame: Day 0 (pre-vaccination), Day 21
Population: PP Set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Quadrivalent VLP Influenza Vaccine - Lot 1 | Quadrivalent VLP Influenza Vaccine - Lot 2 | Quadrivalent VLP Influenza Vaccine - Lot 3
Number analyzed (Participants) | 387 | 383 | 387
percentage of participants
  A/H1N1 (California): Day 0 | 72.3 [67.5 to 76.7] | 76.5 [71.9 to 80.7] | 76.7 [72.2 to 80.9]
  A/H1N1 (California): Day 21 | 96.1 [93.7 to 97.8] | 97.1 [94.9 to 98.6] | 98.7 [97.0 to 99.6]
  A/H3N2 (Hong Kong): Day 0 | 20.0 [16.1 to 24.3] | 19.8 [16.0 to 24.2] | 18.4 [14.6 to 22.6]
  A/H3N2 (Hong Kong): Day 21 | 80.3 [76.0 to 84.2] | 79.6 [75.3 to 83.6] | 77.5 [73.0 to 81.6]
  B/Brisbane: Day 0 | 13.5 [10.2 to 17.3] | 12.3 [9.2 to 16.0] | 13.4 [10.2 to 17.2]
  B/Brisbane: Day 21 | 60.1 [55.0 to 65.0] | 59.8 [54.7 to 64.7] | 55.8 [50.7 to 60.8]
  B/Phuket: Day 0 | 51.6 [46.4 to 56.6] | 58.8 [53.6 to 63.7] | 57.9 [52.8 to 62.9]
  B/Phuket: Day 21 | 90.7 [87.3 to 93.4] | 92.4 [89.3 to 94.9] | 93.8 [90.9 to 96.0]

4. Secondary Outcome: Geometric Mean of the Ratio of GMTs (Geometric Mean Fold Rise [GMFR]) of HI Antibody Response for Each Homologous Influenza Strain
Description: GMFR, the geometric mean of the ratio of GMTs (Day 21/Day 0), was measured using an HI assay for the homologous strains: A/California/7/2009 (H1N1), A/Hong Kong/4801/2014 (H3N2), B/Brisbane/60/2008 (Victoria lineage), and B/Phuket/3073/2013 (Yamagata lineage).
Time Frame: Day 0 (pre-vaccination), Day 21
Population: PP Set.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Quadrivalent VLP Influenza Vaccine - Lot 1 | Quadrivalent VLP Influenza Vaccine - Lot 2 | Quadrivalent VLP Influenza Vaccine - Lot 3
Number analyzed (Participants) | 386 | 383 | 387
ratio
  A/H1N1 (California) | 8.55 [7.66 to 9.53] | 8.43 [7.56 to 9.41] | 8.93 [8.01 to 9.95]
  A/H3N2 (Hong Kong) | 8.41 [7.36 to 9.61] | 8.99 [7.86 to 10.28] | 7.69 [6.73 to 8.78]
  B/Brisbane | 4.08 [3.69 to 4.50] | 4.09 [3.70 to 4.52] | 3.73 [3.38 to 4.12]
  B/Phuket | 5.76 [5.16 to 6.44] | 6.17 [5.53 to 6.90] | 6.30 [5.64 to 7.04]

5. Secondary Outcome: Number of Participants With at Least One Immediate Complaint
Description: Immediate complaints were defined as any solicited local or systemic reactions. Solicited local reactions included: erythema, swelling, and pain at the injection site and solicited systemic reactions included: fever, headache, fatigue, muscle aches, joint aches, chills, a feeling of general discomfort, swelling in the axilla, and swelling in the neck.
Time Frame: 15 minutes post-vaccination
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent VLP Influenza Vaccine - Lot 1 | Quadrivalent VLP Influenza Vaccine - Lot 2 | Quadrivalent VLP Influenza Vaccine - Lot 3
Number analyzed (Participants) | 401 | 398 | 401
Participants | 96 | 108 | 106

6. Secondary Outcome: Number of Participants With at Least One Solicited Local and/or Systemic Reactions
Description: Participants were monitored for both solicited local reactions (erythema, swelling, and pain at the injection site) and solicited systemic reactions (fever, headache, fatigue, muscle aches, joint aches, chills, a feeling of general discomfort, swelling in the axilla, and swelling in the neck). Any solicited local or systemic immediate complaint was also included.
Time Frame: Day 0 (post-vaccination) up to Day 7
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent VLP Influenza Vaccine - Lot 1 | Quadrivalent VLP Influenza Vaccine - Lot 2 | Quadrivalent VLP Influenza Vaccine - Lot 3
Number analyzed (Participants) | 401 | 398 | 401
Participants | 314 | 321 | 321

7. Secondary Outcome: Number of Participants With ≥ Severe Solicited Local and Systemic Reaction
Description: Participants were monitored for both solicited local reactions (erythema, swelling, pain at the injection site) and solicited systemic reactions (fever, headache, fatigue, muscle aches, joint aches, chills, a feeling of general discomfort, swelling in the axilla, swelling in the neck). Any solicited local or systemic immediate complaint was also included. Intensity of solicited reactions graded as mild (1)-easily tolerated and does not interfere with usual activity; moderate (2)-interferes with daily activity, but the participant is still able to function; severe (3)-incapacitating and the participant is unable to work or complete usual activity or potentially life threatening;(4)-likely to be life-threatening if not treated in a timely manner, according to the FDA Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials. The ≥severe events included severe and potentially life-threatening events.
Time Frame: Day 0 (post-vaccination) up to Day 7
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent VLP Influenza Vaccine - Lot 1 | Quadrivalent VLP Influenza Vaccine - Lot 2 | Quadrivalent VLP Influenza Vaccine - Lot 3
Number analyzed (Participants) | 401 | 398 | 401
Participants | 5 | 11 | 6

8. Secondary Outcome: Number of Participants With ≥ Severe Related Solicited Local and Systemic Reactions
Description: Participants were monitored for both solicited local reactions (erythema, swelling, pain at the injection site) and solicited systemic reactions (fever, headache, fatigue, muscle aches, joint aches, chills, a feeling of general discomfort, swelling in the axilla, swelling in the neck). Intensity of solicited reactions was graded according to the FDA toxicity grade: mild (1); moderate (2); severe (3); (4)-likely to be life-threatening if not treated in a timely manner. Causal relationship with study vaccine was assessed as "definitely not related" (clearly not related),"probably not related" (no medical evidence),"possibly related"(reasonable possibility of cause and effect),"probably related"(plausible biologic mechanism and temporal relationship) or "definitely related"(direct cause and effect relationship). The ≥severe events included severe and "potentially life-threatening" and the related category included "possibly related", "probably related", and "definitely related."
Time Frame: Day 0 (post-vaccination) up to Day 7
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent VLP Influenza Vaccine - Lot 1 | Quadrivalent VLP Influenza Vaccine - Lot 2 | Quadrivalent VLP Influenza Vaccine - Lot 3
Number analyzed (Participants) | 401 | 398 | 401
Participants | 3 | 8 | 3

9. Secondary Outcome: Number of Participants With Unsolicited Treatment-Emergent Adverse Events (TEAEs)
Description: Participants were monitored for unsolicited TEAEs. An adverse event (AE) or adverse experience was defined as any untoward medical occurrence in a participant or clinical investigation participant who was administered a pharmaceutical product, with or without a causal relationship with the treatment. An AE can be any favorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to a medicinal product. An AE was considered treatment-emergent if it was aggravated in severity or frequency following the administration of the study vaccine, up to and including the last visit of the study.
Time Frame: Day 0 (post-vaccination) up to Day 21
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent VLP Influenza Vaccine - Lot 1 | Quadrivalent VLP Influenza Vaccine - Lot 2 | Quadrivalent VLP Influenza Vaccine - Lot 3
Number analyzed (Participants) | 401 | 398 | 401
Participants | 94 | 92 | 95

10. Secondary Outcome: Number of Participants With ≥ Severe Unsolicited TEAEs
Description: The intensity of the unsolicited TEAEs was graded as mild (1)-easily tolerated and does not interfere with usual activity; moderate (2)-interferes with daily activity, but the participant is still able to function; severe (3)-incapacitating and the participant is unable to work or complete usual activity or potentially life threatening; (4)-likely to be life-threatening if not treated in a timely manner, according to the FDA Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials. The ≥ Severe events included severe and potentially life-threatening events. AE and TEAEs are defined in outcome measure#9.
Time Frame: Day 0 (post-vaccination) up to Day 21
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent VLP Influenza Vaccine - Lot 1 | Quadrivalent VLP Influenza Vaccine - Lot 2 | Quadrivalent VLP Influenza Vaccine - Lot 3
Number analyzed (Participants) | 401 | 398 | 401
Participants | 4 | 3 | 2

11. Secondary Outcome: Number of Participants With ≥ Severe Related Unsolicited TEAEs
Description: The intensity of the unsolicited TEAEs was graded as: mild (1), moderate (2), severe (3) or potentially life threatening (4). The causal relationship with the study vaccine was assessed as "definitely not related" (clearly not related),"probably not related" (no medical evidence), "possibly related" (reasonable possibility of cause and effect), "probably related" (plausible biologic mechanism and temporal relationship) or "definitely related" (direct cause and effect relationship). The ≥severe events included "severe" and "potentially life-threatening" and the related category included "possibly related", "probably related", and "definitely related." AE and TEAEs are defined in outcome measure #9.
Time Frame: Day 0 (post-vaccination) up to Day 21
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent VLP Influenza Vaccine - Lot 1 | Quadrivalent VLP Influenza Vaccine - Lot 2 | Quadrivalent VLP Influenza Vaccine - Lot 3
Number analyzed (Participants) | 401 | 398 | 401
Participants | 2 | 0 | 0

12. Secondary Outcome: Number of Participants With an Occurrence of Death
Description: The number of participants with an occurrence of death was assessed.
Time Frame: Day 0 (post-vaccination) up to Day 21
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent VLP Influenza Vaccine - Lot 1 | Quadrivalent VLP Influenza Vaccine - Lot 2 | Quadrivalent VLP Influenza Vaccine - Lot 3
Number analyzed (Participants) | 401 | 398 | 401
Participants | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With at Least One Serious TEAE
Description: A serious adverse event (SAE) was considered to be any untoward medical occurrence (whether or not considered to be related to the study vaccine) that, at any dose results in death; is life-threatening (at the time of the event); requires inpatient hospitalization (≥ 24 hours) or prolongation of existing hospitalization (elective hospitalizations/procedures for pre-existing conditions that have not worsened are excluded); results in persistent or significant disability/incapacity; is a congenital abnormality/birth defect; or is another medically important event (e.g. any cases of newly diagnosed cancer). AE and TEAEs is defined in outcome measure #9.
Time Frame: Day 0 (post-vaccination) up to Day 21
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent VLP Influenza Vaccine - Lot 1 | Quadrivalent VLP Influenza Vaccine - Lot 2 | Quadrivalent VLP Influenza Vaccine - Lot 3
Number analyzed (Participants) | 401 | 398 | 401
Participants | 0 | 1 | 0

14. Secondary Outcome: Number of Participants With at Least One AE Leading to Withdrawal
Description: An AE or adverse experience was defined as any untoward medical occurrence in a participant or clinical investigation participant who was administered a pharmaceutical product, with or without a causal relationship with the treatment. An AE can be any favorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to a medicinal product. The number of participants with at least one adverse event leading to withdrawal was assessed.
Time Frame: Day 0 (post-vaccination) up to Day 21
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent VLP Influenza Vaccine - Lot 1 | Quadrivalent VLP Influenza Vaccine - Lot 2 | Quadrivalent VLP Influenza Vaccine - Lot 3
Number analyzed (Participants) | 401 | 398 | 401
Participants | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With at Least One New Onset Chronic Diseases (NOCDs)
Description: All NOCDs that may plausibly have an allergic, autoimmune or inflammatory component were reported. Plausibility should be interpreted broadly; however, the only clear exceptions are degenerative conditions such as osteoarthritis, age-related physiologic changes and life-style diseases. In this context, most cancers, cardiac conditions and kidney diseases should be reported. NOCDs were collected from vaccination on Day 0 to the end of the Day 21 visit.
Time Frame: Day 0 (post-vaccination) up to Day 21
Population: SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent VLP Influenza Vaccine - Lot 1 | Quadrivalent VLP Influenza Vaccine - Lot 2 | Quadrivalent VLP Influenza Vaccine - Lot 3
Number analyzed (Participants) | 401 | 398 | 401
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 0 (post-vaccination) up to 21 days
Description: SAS. The unsolicited SAEs, unsolicited non-serious adverse events (NSAEs), and all deaths were reported.
Arm/Group | Quadrivalent VLP Influenza Vaccine - Lot 1 | Quadrivalent VLP Influenza Vaccine - Lot 2 | Quadrivalent VLP Influenza Vaccine - Lot 3
All-Cause Mortality (participants affected / at risk) | 0/401 | 0/398 | 0/401
Serious Adverse Events (participants affected / at risk) | 0/401 | 1/398 | 0/401
Other Adverse Events (participants affected / at risk) | 94/401 | 92/398 | 95/401
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quadrivalent VLP Influenza Vaccine - Lot 1 (N=401) | Quadrivalent VLP Influenza Vaccine - Lot 2 (N=398) | Quadrivalent VLP Influenza Vaccine - Lot 3 (N=401)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quadrivalent VLP Influenza Vaccine - Lot 1 (N=401) | Quadrivalent VLP Influenza Vaccine - Lot 2 (N=398) | Quadrivalent VLP Influenza Vaccine - Lot 3 (N=401)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gingival abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lymph gland infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 6 (6) | 4 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 15 (15) | 15 (15) | 20 (20)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (2)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Aphonia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 3 (4)
Dizziness exertional (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 11 (14) | 20 (21) | 16 (17)
Migraine (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye swelling (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Neurogenic shock (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 8 (8)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5) | 8 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 (18) | 15 (15) | 8 (9)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) | 3 (3)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (4) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 5 (5) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lip blister (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 7 (7) | 7 (8)
Noninfective gingivitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tongue discolouration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 5 (5) | 3 (3)
Hepatic hypertrophy (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 5 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 3 (3) | 3 (3) | 1 (1)
Urachal abnormality (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 1 (1)
Discomfort (General disorders) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 4 (4) | 6 (6) | 4 (4)
Hangover (General disorders) | 1 (1) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 2 (2) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 1 (1) | 1 (1) | 1 (1)
Injection site irritation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site joint discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site warmth (General disorders) | 0 (0) | 1 (1) | 3 (3)
Local swelling (General disorders) | 1 (1) | 2 (2) | 2 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 2 (2)
Vaccination site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Superficial injury of eye (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator understands that the information in the protocol is confidential and should not be disclosed, other than to those directly involved in the execution or the ethical review of the study, without prior written authorization from the Sponsor. It is, however, permissible to discuss information contained in the protocol with a participant in order to obtain consent once Institutional Review Board (IRB) approval is obtained.

DOCUMENTS (2):
  • Study Protocol (2017-08-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT03321968/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT03321968/SAP_001.pdf